CLINICAL TRIAL: NCT06676033
Title: Correlative Study of Epcoritamab in Chronic Lymphocytic Leukemia and Richter Syndrome
Brief Title: Epcoritamab in Chronic Lymphocytic Leukemia and Richter Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10001671; 001671-H
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10-03

CONDITIONS: Leukemia, Chronic Lymphocytic; Richter Syndrome
Keywords: Epcoritamab, Pharmacodynamic, Tumor Microenvironment, Clonal Dynamics, Biomarker
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- epcoritamab (Experimental): Samples from subjects receiving epcoritamab on another clinical trial GCT3013-03 will be collected.
  Interventions: Drug: epcoritamab

INTERVENTIONS:
Drug: epcoritamab — Samples from subjects receiving epcoritamab on another clinical trial GCT3013-03 will be collected.

SUMMARY:
This correlative study aims to understand the pharmacodynamic effects and clonal dynamics in response to epcoritamab by obtaining and analyzing lymph node, bone marrow, and blood samples from subjects enrolled in GCT3013-03 trial sponsored by Genmab at NIH. Samples will be collected before and at multiple time points during treatment with epcoritamab. National Heart, Lung, and Blood Institute (NHLBI) investigators are experienced in testing samples treated with bsAb2,3 including epcoritamab in an ongoing pre-clinical collaboration with Genmab. Addressing the objectives of this correlative study will advance the science and clinical application of epcoritamab specifically as well as T-cell engaging bsAb in general as an emerging class of immunotherapy for cancer.

The study is enrolling by invitation only.

DETAILED DESCRIPTION:
Study Description:

Subjects enrolled in GCT3013-03, a phase 1b/2 study of epcoritamab in R/R CLL and RS, at the National Institutes of Health (NIH) Clinical Center (CC) will be invited to simultaneously participate in this companion correlative study. Subjects will undergo percutaneous lymph node coreneedle biopsies, bone marrow biopsies, lymphapheresis, and blood draws for pharmacodynamic evaluation of tumor and immune cells in affected tissue sites and blood before and during treatment with epcoritamab.

Objectives:

Primary Objective:

-Assess the pharmacodynamic effects of epcoritamab in the tumor microenvironment.

Secondary Objectives:

* Assess the pharmacodynamic effects of epcoritamab in blood
* Investigate clonal dynamics during treatment with epcoritamab

Exploratory Objective:

-Evaluate pharmacodynamic and predictive biomarkers

Endpoints:

Primary Endpoint:

-Immunophenotype and transcriptome of T cells and tumor cells in lymph node and bone marrow

Secondary Endpoints:

* Immunophenotype and transcriptome of T cells and tumor cells in peripheral blood
* DNA sequencing of tumor cells

Exploratory Endpoints:

-Tests include, but are not limited to single cell multiomics, bulk lymph node transcriptome cytokine analysis

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Must be undergoing screening for GCT3013-03
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Immunophenotype and transcriptome of T cells and tumor cells in lymph node and bone marrow | 25 days (Cycle 1 Day 25)

SECONDARY OUTCOMES:
Immunophenotype and transcriptome of T cells and tumor cells in peripheral blood | 167 Days (Cycle 7 Day 1)
DNA sequencing of tumor cells | 167 Days (Cycle 7 Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian U Wiestner, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The clinical components of this project will generate data as specified by the clinical protocols, including patient demographics, tumor characteristics, treatment administration, and response, adverse events, and other primary/secondary outcomes. Data will be collected from all enrolled research participants. To protect research participant identities, individual de-identified data points will be made available for sharing. protocol-related clinical data as generated above will be preserved as specified by the clinical protocol. Shared data will be limited to that specified within the protocol informed consent. Shared data will be aggregated as necessary to ensure deidentification of the data in accordance with applicable legal and regulatory requirements governing human subjects' research.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by the end of the project/protocol or at the time of associated publication, whichever comes first.
Access Criteria: BioData Catalyst is supported by NHLBI and access to data is controlled by the NHLBI Data Access Committee (DAC) utilizing the database of Genotypes and Phenotypes (dbGaP) permissions infrastructure. In order to access controlled-access data in BioData Catalyst, an investigator must have an approved Data Access Request (DAR) in dbGaP.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001671-H.html